CLINICAL TRIAL: NCT01998750
Title: Study to Identify Rare Genetic Variants Causing Severe Early Childhood Obesity
Brief Title: Study to Investigate Genetic Causes of Severe Early Childhood Onset Obesity.
Acronym: GECO
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Boston Children's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Vidhu V. Thaker, Assistant Professor, Columbia University
Other Study IDs: AAAR0351; P00009351 (Other: Boston Children's Hospital); 5K23DK110539-03 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: obesity; genetics; early-onset; childhood
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early-onset severe obesity: The study will enroll individuals with early onset severe obesity (BMI > 99th percentile noted at an age < 6 years of age). Individuals with a known history of early onset obesity are eligible, regardless of their current age.

SUMMARY:
This study aims to investigate genetic causes of early childhood obesity.

The investigators will enroll children and adults with severe early onset obesity (BMI > 99th percentile) diagnosed prior to 6 years of age. The investigators will ask questions about the health and eating behavior of the participants, and perform a brief physical examination. The investigators will collect saliva or blood to perform genetic testing from the participants and invite family members to enroll in the study.

DETAILED DESCRIPTION:
This is a clinical and genomic study designed to investigate monogenic causes of severe early childhood obesity.

Participants with severe early onset obesity will be identified by screening of the clinical database or referred for the study. These subjects will be invited to participate in the study. After obtaining informed consent, the investigators will obtain history on the proband and the family, and perform a brief examination in addition to collecting genetic material.

Targeted sequencing of genes associated with monogenic and syndromic forms of obesity will be performed using next-generation sequencing. In selected individuals with favorable family history, exome or whole genome sequencing will be performed. Functional analysis of newly identified variants will be performed where possible.

ELIGIBILITY:
Inclusion Criteria:

- BMI > 99th percentile documented at age < 6 years of age

Exclusion Criteria:

* Known genetic causes of obesity
* Known Endocrine causes of obesity.
* Neurologic tumor, trauma or surgery
* Prior malignancy or transplant
* Known autoimmune diseases
* Edema of a known or unknown cause
* Prolonged steroid use.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll children with BMI > 99th percentile for age noted prior to 6 years of age. Current age of the child can vary from 0-21 years.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-02; Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of known or novel genetic variants in genes that underlie obesity. | 1.5-2 years
  Identification of known or novel genetic variants in genes that underlie obesity.

SECONDARY OUTCOMES:
Prevalence of melanocortin receptor 4 mutations. | 2 years
  We will test the hypothesis that 1-3% of early onset obesity could be explained by carriage of mutation of monogenic obesity such as melanocortin receptor 4 in a mixed pediatric population.

CONTACTS AND LOCATIONS:
Overall Officials: Vidhu Thaker, M.D., Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be deposited in public databases at the end of the study

REFERENCES:
- [Result] De Rosa MC, Chesi A, McCormack S, Zhou J, Weaver B, McDonald M, Christensen S, Liimatta K, Rosenbaum M, Hakonarson H, Doege CA, Grant SFA, Hirschhorn JN, Thaker VV. Characterization of Rare Variants in MC4R in African American and Latino Children With Severe Early-Onset Obesity. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2961-2970. doi: 10.1210/jc.2018-02657. PMID 30811542